CLINICAL TRIAL: NCT07063030
Title: An Exploratory Clinical Study to Evaluate LX107 Gene Therapy in Patients With AIPL1 Biallelic Mutation-related Inherited Retinal Dystrophy (AIPL1-IRD)
Brief Title: A Study of LX107 Gene Therapy in AIPL1-IRD Patients
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Collaborators: Innostellar Biotherapeutics Co.,Ltd (Industry)
Responsible Party: Principal Investigator, Xiaodong Sun, Director, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHGH-LX107
Record Dates: First submitted 2025-07-03; First posted 2025-07-14 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Retinal Dystrophy
MeSH Terms: conditions — Retinal Dystrophies

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Experimental: LX107 Injection
  Arm Description:
  * Low dose group: subretinal injection of LX107 -3×10⁹ VG/eye
  * Medium dose group: subretinal injection of LX107- 1×10¹⁰ VG/eye
  * High dose group: subretinal injection of LX107 -3×10¹⁰ VG/eye
  Interventions: Genetic: LX107 Injection

INTERVENTIONS:
Genetic: LX107 Injection — Subjects will receive subretinal injection of LX107 on Day 0.

SUMMARY:
Administering subretinal injection of LX107 injection (a gene therapy drug) to patients with retinal dystrophy caused by AIPL1 gene mutation to evaluate its efficacy and safety.

ELIGIBILITY:
Inclusion Criteria:

1. The subject and/or their guardian signs a written informed consent form and is willing to comply with the long-term follow-up protocol and supporting protocols.
2. Adult or pediatric patients (aged ≥ 4 years) diagnosed with AIPL1-IRD.
3. Definitive molecular diagnosis of biallelic AIPL1 gene mutations confirmed by next-generation sequencing combined with Sanger validation.
4. The study eye has a best-corrected visual acuity of no more than 58 letters (approximately equivalent to decimal visual acuity ≤ 0.3) using the ETDRS visual acuity chart at baseline.

Note: Only one eye will be designated as the "study eye" (i.e., the eye to receive treatment) at the investigator's discretion.

Exclusion Criteria:For any eye with the following conditions:

1. A history of ocular diseases that, in the investigator's judgment, may hinder the planned treatment or interfere with the interpretation of study endpoints (e.g., glaucoma, diabetic retinopathy, retinal vein occlusion, retinal detachment, posterior or panuveitis, etc.).
2. Any eye with a history of gene therapy for IRD or other hereditary neuro-ophthalmic diseases (including but not limited to other viral vector-based gene therapies, mRNA therapies, etc.).
3. A lack of sufficient viable retinal cells as determined by non-invasive methods such as OCT or ophthalmoscopy.
4. Any active intraocular or periocular infection in the study eye (e.g., infectious conjunctivitis, keratitis, scleritis, endophthalmitis, infectious blepharitis, uveitis).
5. A history of intraocular surgery (e.g., vitrectomy, cataract surgery, trabeculectomy, or other filtering surgery) in the 6 months prior to the screening visit.

   For any systemic conditions:
6. Uncontrolled hypertension, defined as systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg. If the initial measurement exceeds the above limits, it may be repeated on the same day or another day during the screening period; if the subject is taking oral antihypertensive drugs, they must have been on a stable dose of the same drug for at least 30 days prior to screening.
7. Diabetic patients meeting any of the following criteria: ① known to have macrovascular complications; ② baseline HbA1c > 7.5%; ③ receiving treatment with two or more oral hypoglycemic agents, insulin, or GLP-1 receptor agonists.
8. A history of any other diseases, metabolic disorders, physical examination findings, or clinical laboratory abnormalities that, in the investigator's judgment, may contraindicate the use of the study drug, interfere with the interpretation of study results, or place the subject at high risk of treatment complications, including but not limited to: AIDS, syphilis, acute/chronic active hepatitis B or C, coagulation disorders, a history of treated or untreated malignancy within the past 5 years (except for localized basal cell carcinoma of the skin or in situ cervical cancer), etc.
9. Any of the following laboratory abnormalities: ① platelet count < 100 × 10⁹/L, hemoglobin (Hb) < 10 g/dL (males) or < 9 g/dL (females); ② aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 3 × ULN; ③ serum creatinine or urea > 1.5 × ULN.
10. Administration of any other investigational drug (except vitamins and minerals) within 3 months prior to screening, or an attempt to participate in another clinical trial during the study period.
11. Other circumstances deemed unsuitable for enrollment by the investigator.
12. Unwillingness to use effective contraceptive methods during the study; pregnant or lactating women, or women planning to become pregnant or lactate during the study period.

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 6 Months
  Incidence of ocular and non-ocular adverse events (AEs) and serious adverse events (SAEs) following LX107 subretinal injection

SECONDARY OUTCOMES:
Changes in Functional Magnetic Resonance Imaging (fMRI) Results | 6 months、12 months
Mean Change from Baseline in Multi-luminance Mobility Test (MLMT) | 6 months、12 months
  Assess the subject's mobility ability under different light intensities using MLMT, and compare the mean changes from baseline at 180 and 365 days after treatment to reflect improvements in visual function.
Mean Change from Baseline in Full-Field Sensitivity Threshold (FST) | 6 months、12 months
  Measure the subject's light perception ability using FST, and compare the mean changes from baseline at 180 and 365 days after treatment to evaluate improvements in visual sensitivity.
Mean Change from Baseline in Visual Acuity (VA) | 6 months、12 months
  Measure VA using ETDRS and BRVT charts, with LogMAR score as the indicator, and compare the mean changes from baseline at 180 and 365 days after treatment to assess visual acuity improvement.
Mean Change from Baseline in Visual Fields | 6 months、12 months
  Use Goldmann perimeter (dynamic visual field) and Humphrey perimeter (static visual field) to compare the mean changes from baseline at 180 and 365 days after treatment, evaluating improvements in visual field range and sensitivity.

IPD SHARING:
Plan to Share IPD: No